CLINICAL TRIAL: NCT01325779
Title: Prevention of Lower Extremity Deep Venous Thrombosis in the Surgical Intensive Care Unit: a Randomized Trial Comparing Subcutaneous Heparin and Subcutaneous Enoxaparin
Brief Title: Comparison of Subcutaneous Heparin and Enoxaparin for Deep Venous Thrombosis (DVT) Prophylaxis in Surgical Intensive Care Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Lisa Louwers (Other)
Responsible Party: Sponsor-Investigator, Lisa Louwers, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HIC 2010-113
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Lower Extremity Deep Venous Thrombosis
Keywords: deep venous thrombosis; DVT; enoxaparin; heparin; surgical intensive care
MeSH Terms: conditions — Venous Thrombosis | interventions — Heparin; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- subcutaneous heparin (Active Comparator)
  Interventions: Drug: heparin
- subcutaneous enoxaparin (Active Comparator)
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: heparin — subcutaneous heparin 5000 units every 8 hours
  Arms: subcutaneous heparin
Drug: enoxaparin — subcutaneous enoxaparin 40 milligrams every 24 hours
  Arms: subcutaneous enoxaparin

SUMMARY:
Study hypothesis: Subcutaneous enoxaparin is more effective than subcutaneous heparin in preventing the development of DVT in the general surgical intensive care unit population.

Hospitalized patients are at increased risk for the development of blood clots in the legs, known as deep venous thrombosis (DVT). Surgical patients are in a higher risk category than the general hospital population due to a number of factors including undergoing surgery and increased risk of immobility. The highest risk patients are in the surgical intensive care unit, where their surgical risks for blood clots are combined with issues such as sepsis, acquired blood clotting disorders, and increasing age, each of which are factors that contribute to the risk of blood clot development. 1. Patients who develop these blood clots (DVTs) are at risk for chronic leg swelling, pain, and in some cases, chronic ulcer development on the leg. In the worst case scenario, these blood clots can break away and migrate to the lungs where they cause a pulmonary embolism (PE), a clot in the lungs that can cause significant breathing difficulty requiring intubation and mechanical ventilation, and in some cases, death.

According to recent research, DVTs account for over 200,000 patient deaths each year nationwide. 2. A large amount of data has supported the use of medication called heparin or enoxaparin in low doses to prevent these blood clots from forming while in the hospital. Both of these medications are considered standard of care for use patients considered moderate and high risk for the development of DVT. 3. While both of these medications have been shown to significantly reduce the occurrence of DVT in appropriate doses, 4. there has never been a direct comparison of the two medications in the highest-risk population of the surgical intensive care unit. Our own preliminary data suggests patients may have a lower incidence of DVTs with the use of enoxaparin versus heparin. Part of the reason for this may be the requirement for three times daily dosing of the heparin compared to once daily dosing for enoxaparin. There may also be some inherent differences in the efficacy of the medications themselves.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* admission to the surgical intensive care unit
* admitting physician is a surgeon or patient is status-post a surgical procedure

Exclusion Criteria:

* age < 18 years old
* inability to obtain informed consent from patient or legal representative within 24 hours of SICU admission
* patient admitted to neurosurgery or status-post a neurosurgical procedure
* patient status-post an orthopedic procedure
* patient admitted with a primary diagnosis of trauma
* patient with a history of a bleeding disorder or other contraindication to even low-dose anticoagulation medicine including a history of heparin-induced thrombocytopenia verified with a positive serotonin-release assay or have a high clinical suspicion of new onset heparin-induced thrombocytopenia resulting in the discontinuation of heparin or enoxaparin by the treating physicians
* patients on current full anticoagulation medications including a heparin drip or warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Development of lower extremity deep venous thrombosis | hospital admission (day 1 ) to 3 months post discharge

SECONDARY OUTCOMES:
Adverse events associated with use of subcutaneous heparin and enoxaparin | hospital admission (day 1) through discharge

CONTACTS AND LOCATIONS:
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States